CLINICAL TRIAL: NCT04677621
Title: Telemedicine Nurse DBS for Parkinson's Disease: The TEND Study
Brief Title: TEND Study:Telemedicine Nurse DBS for Parkinson's Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding never received closed with the IRB
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB202002994-N; OCR39945 (Other: UF OnCore); PRO00042966 (Other: UFIRST)
Record Dates: First submitted 2020-12-17; First posted 2020-12-21 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Parkinson Disease
Keywords: Home Health
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse Telehealth Intervention (Experimental): Allocated to tele-intervention
  Interventions: Other: Nurse Telehealth
- Standard Deep Brain Stimulation (DBS) (Active Comparator): Allocated to conventional approach
  Interventions: Other: STANDARD DBS

INTERVENTIONS:
Other: Nurse Telehealth — Subjects will receive nurse telehealth Mobile Decision Support System (MAP) DBS care
  Arms: Nurse Telehealth Intervention
Other: STANDARD DBS — Subjects will receive standard in-person clinic-based DBS care administered without the use of Mobile Decision Support System (MAP) DBS
  Arms: Standard Deep Brain Stimulation (DBS)

SUMMARY:
The central hypothesis is that home health nurses can improve access and provide high quality care when guided by a sophisticated platform that integrates bioinformatics, patient-specific computational modeling, and continuous symptom measurement.

ELIGIBILITY:
Inclusion Criteria:

* Pre-operative Inclusion Criteria: A good response to levodopa is required in order to exclude patients with Parkinson's plus syndromes, and will be defined as a 30% improvement in parkinsonian motor signs based upon the Unified PD Rating Scale (UPDRS) motor examination subscore, following the administration of 1.5 times the typical dopaminergic dose during the screening neurological examination. Patients must also have PD for a minimum of 5 years duration.
* Additional inclusion criteria consist of: 1) Hoehn & Yahr stage II or worse when off; 2) Intractable, disabling motor fluctuations and/or tremor; 3) Age between 30-75 years; 4) Unsatisfactory clinical response to maximal medical management (with trials of both higher and lower doses of antiparkinsonian drugs). 5) A stable/optimal medical regimen of antiparkinsonian drug therapy for at least one month prior to surgery; 6) access to high-speed internet in the home.

Exclusion Criteria:

* Clinically significant medical disease that would increase the risk of developing pre- or postoperative complications (e.g. significant cardiac or pulmonary disease, uncontrolled hypertension).
* Evidence of secondary or atypical parkinsonism.
* MRI scan with significant evidence of brain atrophy or other abnormalities.
* Dementia as evidenced by impairment in two neuropsychological domains and impaired or borderline neuropsychological function in one additional domain.
* A major untreated psychiatric disorder.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
The number of participant clinic visits | 6 MONTHS from date of enrollment
  The number of in-person clinic visits required for each participant during the 6-month post operative DBS period.

SECONDARY OUTCOMES:
PDQ-39 Scores | 6-months
  Difference in PDQ-39 scores from baseline to the 6-month time point. PDQ summary index score 0-very good to 100 bad

OTHER OUTCOMES:
UPDRS scores | 6-months
  Difference in UPDRS scores from baseline to 6-month time point. UPDRS scoring scale 0-very good to 100-bad

CONTACTS AND LOCATIONS:
Overall Officials: Michael Okun, MD, Principal Investigator — University of Florida

IPD SHARING:
Plan to Share IPD: No